CLINICAL TRIAL: NCT01493037
Title: Pressure Controlled Intermittent Coronary Sinus Occlusion in Patients With ST Segment Elevation Myocardial Infarction Treated by Primary Percutaneous Coronary Intervention: Safety and Feasibility Study
Brief Title: PICSO in Patients With STEMI Treated by Primary Percutaneous Coronary Intervention
Acronym: pRAMSES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miracor Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP 2011-01
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction
Keywords: STEMI; PICSO; Coronary Sinus; Involving Left Anterior Descending Coronary Artery
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PICSO (Other): PICSO treatment for 90 minutes
  Interventions: Device: PICSO (Pressure-controlled Intermittent Coronary Occlusion

INTERVENTIONS:
Device: PICSO (Pressure-controlled Intermittent Coronary Occlusion — The PICSO catheter has a balloon which is placed in the coronary sinus via the femoral vein. The balloon is inflated and deflated at intervals calculated by an algorithm and adjusted according to the patient's own coronary sinus pressure plateau.
  Other Names: PICSO Impulse Catheter; PICSO Impulse Console

SUMMARY:
A prospective multi-center study in which patients with an acute heart attack (in the left anterior descending artery) with ECG changes (ST segment elevation) receive angioplasty followed by stent placement and 90 minutes of PICSO treatment. This is a proof of concept study designed to document the safety and feasibility of the Pressure Controlled Intermittent Coronary Sinus Occlusion (PICSO) Impulse system.

ELIGIBILITY:
Inclusion Criteria:

* First time anterior STEMI defined by the following:

  * Symptoms of myocardial ischemia > 30 minutes and < 12 hours
  * ST-segment elevation > 1mm (> 0.1 mV) in two contiguous precordial leads in the anterior territory on a 12-lead ECG
* Uncomplicated PCI of a LAD culprit lesion (defined as angioplasty followed by stent placement or direct stenting without the occurrence of an adverse event(s) that would preclude further study participation, such as major bleeding, perforation, hypotension, pulmonary edema or instability that in the judgement of the investigator preclude participation in the trial)

Exclusion Criteria:

* Younger than 18 years of age
* Hospitalization with a primary diagnosis of acute myocardial infarction (AMI) previously or has evidence of previous Q-wave infarct
* Left main coronary artery culprit lesion
* Additional stenosis in the LAD for which PCI or CABG is likely to be needed in the next 6 months and which is not treated during the index procedure
* Cardiogenic shock (systolic blood pressure ≤90 mmHg in spite of conservative measures) or pulmonary edema (O2 saturation <90% by pulse oximetry and the presence of rales or crackles)
* Cardiac arrest requiring chest compression or resuscitation
* Anatomical complications limit capacity to place PICSO Impulse device or achieve stable catheter placement or occlude coronary sinus
* Known renal disease (GFR < 30 mL/min/1.73m2) or dialysis
* History of stroke, TIA or reversible ischemic neurological disease within last 6 months
* Left bundle branch block
* Known contra-indication for magnetic resonance imaging (Metallic implant precluding MRI, claustrophobia, obesity precluding MRI, etc.)
* Presence of any lead in the coronary sinus
* Active or treated malignancies in the last 12 months
* Previous coronary artery bypass graft surgery
* Known severe anemia (Hgb < 10 g/dL or < 6.2 mmol/L)
* Known platelet count < 100,000, known coagulopathy or bleeding diathesis, or unwilling to accept transfusions
* Participation in another ongoing clinical study
* Women of child-bearing age
* Non-cardiac comorbidities and life expectancy < 1 year
* Legal incompetence
* A condition that, in the opinion of the Investigator, precludes participation, including compliance with all follow-up procedures
* No dependents neither to the sponsor nor to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Successful delivery of PICSO treatment | 90 minutes
  Assessment of the feasibiity of PICSO in STEMI patients defined as the successful elivery of the PICSO catheter and the successful administration of PICSO treatment for 90 minutes

SECONDARY OUTCOMES:
MRI measurement of infarct size | 4 months
  Infarct size assessed by cardiac MRI between 2-5 days post primary PCI and again at 120 days follow up
Assessment of left ventricular function | 4 months
  Left ventricular function assessed by echocardiography between 2-5 days after primary PCI and at 120 days
Assessment of microvascular perfusion | 4 months
  Microvascular perfusion assessed by cardiac MRI between 2-5 days after primary PCI and at 120 days
Resolution of ST-segment elevation | 24 hours
  Occurrence of complete resolution of ST-segment elevation 30, 60, 90 and 120 minutes after last contrast injection prior to PICSO placement procedure on 24 hour continuous 12 lead ECG Holter monitor recording
Measurement of ST segment time curve area | 3 hours
  ST segment time curve area for the first 3 hours on 24 hour continuous 12 lead ECG Holter monitor recording.
Number of adverse events | 6 months
  Safety endpoints recorded are Major Adverse Cardiac Events (MACE), Major Adverse Cardiac and Cerebrovascular Events (MACCE), net adverse clinical events (MACE and bleeding), Serious and non serious Adverse Device Events ((S)ADE) rates

CONTACTS AND LOCATIONS:
Overall Officials: Jan J Piek, Professor, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Academic Medical Center - University of Amsterdam, Amsterdam
  - Amphia Hospital, Breda